CLINICAL TRIAL: NCT00007761
Title: CSP #430 - Reducing The Efficacy-Effectiveness Gap In Bipolar Disorder
Brief Title: Does Bipolar Disease Program (BDP) Intervention Improve Long Term Manic and Depressive Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bauer, Mark - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 430
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disease Program intervention
MeSH Terms: conditions — Bipolar Disorder | interventions — Psychiatry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bipolar Disorder Program
  Interventions: Behavioral: Bipolar Disorder Program
- 2 (Active Comparator): Usual (psychiatric) Care
  Interventions: Behavioral: Usual (psychiatric) Care

INTERVENTIONS:
Behavioral: Bipolar Disorder Program
  Arms: 1
Behavioral: Usual (psychiatric) Care
  Arms: 2

SUMMARY:
Based on highly promising preliminary data, it is proposed to conduct a multi-site randomized controlled trial of a high-intensity ambulatory treatment program for bipolar disorder against standard office-based, physician-centered care. The major characteristics of this program are that it emphasizes (1) aggressive guideline-driven pharmacotherapy, (2) continuity of care with identified primary mental health nurse clinicians supported by psychiatrist back-up, and (3) patient education to improve treatment alliance and illness management skills.

DETAILED DESCRIPTION:
Primary Hypothesis: The primary hypotheses are that Bipolar Disease Program (BDP) intervention will significantly improve (1) manic and (2) depressive symptom scores, as well as Total Treatment Costs as compared to usual care of bipolar patients.

Secondary Hypothesis: Secondary hypotheses include significant improvement in BDP patients as compared to usual bipolar treatment care with respect to functional outcome, quality of life, intensity of somatotherapy, patient satisfaction, and provider attitudes.

Intervention: Usual (psychiatric) Care vs Bipolar Disorder Program

Primary Outcomes: The primary outcomes are: (1) Manic Symptom Score; (2) Depressive Symptom Score; and (3) Total Treatment Costs.

Study Abstract: Based on highly promising preliminary data, it is proposed to conduct a multi-site randomized controlled trial of a high-intensity ambulatory treatment program for bipolar disorder against standard office-based, physician-centered care. The major characteristics of this program are that it emphasizes (1) aggressive guideline-driven pharmacotherapy, (2) continuity of care with identified primary mental health nurse clinicians supported by psychiatrist back-up, and (3) patient education to improve treatment alliance and illness management skills.

Patients with bipolar disorder will be randomly assigned to either standard care or the high intensity ambulatory program for three years. Outcome variables will cover three distinct domains: disease-specific outcome (number, length, and severity of manic and depressive episodes), functional outcome (social and occupational role function and subjective quality of life), and total treatment costs (direct treatment costs and indirect costs of illness). Preliminary data indicate that these domains are related but not redundant. Each of these is relevant to patient well-being and to VHA management.

ELIGIBILITY:
Inclusion Criteria:

Patients with bipolar disorder. Index episode of manic, major depression or both requiring hospitalization on acute unit. At lease two hospitalizations, three or more months apart within the past 5 years.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 1997-07; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Bauer, MD BA, Study Chair — VA Boston Healthcare System, Brockton Campus
Locations (13):
- United States (13):
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Augusta, Augusta, Georgia
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - James H. Quillen VA Medical Center, Mountain Home, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas

REFERENCES:
- [Result] Pirraglia PA, Biswas K, Kilbourne AM, Fenn H, Bauer MS. A prospective study of the impact of comorbid medical disease on bipolar disorder outcomes. J Affect Disord. 2009 Jun;115(3):355-9. doi: 10.1016/j.jad.2008.09.020. Epub 2008 Oct 18. PMID 18930558
- [Result] Brown GR, McBride L, Bauer MS, Williford WO; Cooperative Studies Program 430 Study Team. Impact of childhood abuse on the course of bipolar disorder: a replication study in U.S. veterans. J Affect Disord. 2005 Dec;89(1-3):57-67. doi: 10.1016/j.jad.2005.06.012. Epub 2005 Oct 4. PMID 16213029
- [Result] Bauer MS, Williford WO, McBride L, McBride K, Shea NM. Perceived barriers to health care access in a treated population. Int J Psychiatry Med. 2005;35(1):13-26. doi: 10.2190/U1D5-8B1D-UW69-U1Y4. PMID 15977942
- [Result] Bauer MS, Altshuler L, Evans DR, Beresford T, Williford WO, Hauger R; VA Cooperative Study #430 Team. Prevalence and distinct correlates of anxiety, substance, and combined comorbidity in a multi-site public sector sample with bipolar disorder. J Affect Disord. 2005 Apr;85(3):301-15. doi: 10.1016/j.jad.2004.11.009. PMID 15780700
- [Result] Bauer MS, Mitchner L. What is a "mood stabilizer"? An evidence-based response. Am J Psychiatry. 2004 Jan;161(1):3-18. doi: 10.1176/appi.ajp.161.1.3. PMID 14702242
- [Result] Glick HA, McBride L, Bauer MS. A manic-depressive symptom self-report in optical scanable format. Bipolar Disord. 2003 Oct;5(5):366-9. doi: 10.1034/j.1399-5618.2003.00043.x. PMID 14525558
- [Result] Bauer MS. An evidence-based review of psychosocial treatments for bipolar disorder. Psychopharmacol Bull. 2001 Summer;35(3):109-34. PMID 12397882
- [Result] Bauer MS. A review of quantitative studies of adherence to mental health clinical practice guidelines. Harv Rev Psychiatry. 2002 May-Jun;10(3):138-53. doi: 10.1080/10673220216217. PMID 12023929
- [Result] Bauer MS. The collaborative practice model for bipolar disorder: design and implementation in a multi-site randomized controlled trial. Bipolar Disord. 2001 Oct;3(5):233-44. doi: 10.1034/j.1399-5618.2001.30502.x. PMID 11903206
- [Result] Bauer MS, Kirk GF, Gavin C, Williford WO. Determinants of functional outcome and healthcare costs in bipolar disorder: a high-intensity follow-up study. J Affect Disord. 2001 Aug;65(3):231-41. doi: 10.1016/s0165-0327(00)00247-0. PMID 11511403
- [Result] Vojta C, Kinosian B, Glick H, Altshuler L, Bauer MS. Self-reported quality of life across mood states in bipolar disorder. Compr Psychiatry. 2001 May-Jun;42(3):190-5. doi: 10.1053/comp.2001.23143. PMID 11349236
- [Result] Bauer MS, Vojta C, Kinosian B, Altshuler L, Glick H. The Internal State Scale: replication of its discriminating abilities in a multisite, public sector sample. Bipolar Disord. 2000 Dec;2(4):340-6. doi: 10.1034/j.1399-5618.2000.020409.x. PMID 11252648
- [Result] Sajatovic M, Biswas K, Kilbourne AK, Fenn H, Williford W, Bauer MS. Factors associated with prospective long-term treatment adherence among individuals with bipolar disorder. Psychiatr Serv. 2008 Jul;59(7):753-9. doi: 10.1176/ps.2008.59.7.753. PMID 18586992
- [Result] Altshuler L, Tekell J, Biswas K, Kilbourne AM, Evans D, Tang D, Bauer MS. Executive function and employment status among veterans with bipolar disorder. Psychiatr Serv. 2007 Nov;58(11):1441-7. doi: 10.1176/ps.2007.58.11.1441. PMID 17978254
- [Result] Bauer MS, McBride L, Williford WO, Glick H, Kinosian B, Altshuler L, Beresford T, Kilbourne AM, Sajatovic M; Cooperative Studies Program 430 Study Team. Collaborative care for bipolar disorder: Part II. Impact on clinical outcome, function, and costs. Psychiatr Serv. 2006 Jul;57(7):937-45. doi: 10.1176/ps.2006.57.7.937. PMID 16816277
- [Result] Bauer MS, McBride L, Williford WO, Glick H, Kinosian B, Altshuler L, Beresford T, Kilbourne AM, Sajatovic M; Cooperative Studies Program 430 Study Team. Collaborative care for bipolar disorder: part I. Intervention and implementation in a randomized effectiveness trial. Psychiatr Serv. 2006 Jul;57(7):927-36. doi: 10.1176/ps.2006.57.7.927. PMID 16816276
- [Result] Sajatovic M, Bauer MS, Kilbourne AM, Vertrees JE, Williford W. Self-reported medication treatment adherence among veterans with bipolar disorder. Psychiatr Serv. 2006 Jan;57(1):56-62. doi: 10.1176/appi.ps.57.1.56. PMID 16399963
- [Result] Fenn HH, Bauer MS, Altshuler L, Evans DR, Williford WO, Kilbourne AM, Beresford TP, Kirk G, Stedman M, Fiore L; VA Cooperative Study #430 Team. Medical comorbidity and health-related quality of life in bipolar disorder across the adult age span. J Affect Disord. 2005 May;86(1):47-60. doi: 10.1016/j.jad.2004.12.006. PMID 15820270
- [Result] Kilbourne AM, Bauer MS, Pincus H, Williford WO, Kirk GF, Beresford T; Veterans Administration (VA) Cooperative Study #430 Team. Clinical, psychosocial, and treatment differences in minority patients with bipolar disorder. Bipolar Disord. 2005 Feb;7(1):89-97. doi: 10.1111/j.1399-5618.2004.00161.x. PMID 15654937
- [Result] Glick HA, Kinosian B, McBride L, Williford WO, Bauer MS; CSP #430 Study Team. Clinical nurse specialist care managers' time commitments in a disease-management program for bipolar disorder. Bipolar Disord. 2004 Dec;6(6):452-9. doi: 10.1111/j.1399-5618.2004.00159.x. PMID 15541060
- [Result] Polsky D, Onesirosan P, Bauer MS, Glick HA. Duration of therapy and health care costs of fluoxetine, paroxetine, and sertraline in 6 health plans. J Clin Psychiatry. 2002 Feb;63(2):156-64. doi: 10.4088/jcp.v63n0212. PMID 11874218
- [Result] Bauer MS, Williford WO, Dawson EE, Akiskal HS, Altshuler L, Fye C, Gelenberg A, Glick H, Kinosian B, Sajatovic M. Principles of effectiveness trials and their implementation in VA Cooperative Study #430: 'Reducing the efficacy-effectiveness gap in bipolar disorder'. J Affect Disord. 2001 Dec;67(1-3):61-78. doi: 10.1016/s0165-0327(01)00440-2. PMID 11869753
- [Result] Kilbourne AM, Biswas K, Pirraglia PA, Sajatovic M, Williford WO, Bauer MS. Is the collaborative chronic care model effective for patients with bipolar disorder and co-occurring conditions? J Affect Disord. 2009 Jan;112(1-3):256-61. doi: 10.1016/j.jad.2008.04.010. Epub 2008 May 27. PMID 18504059